CLINICAL TRIAL: NCT05776875
Title: Atezolizumab and Bevacizumab in Combination With TACE for Patients With BCLC B HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000026840; 000 (Other: CTGTY)
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma; BCLC Stage B Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm study which will be performed to examine the safety and tolerability of the combination of atezolizumab and bevacizumab with TACE for patients with BCLC B HCC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab and Bevacizumab in combination with TACE (Experimental): THIS IS A SINGLE ARM PILOT/FEASABILITY STUDY. THE STUDY CONSISTS OF A SCREENING PERIOD (DAY -28 TO DAY -1), A TREATMENT PERIOD, AND A TREATMENT DISCONTINUATION VISIT.
  The atezolizumab and bevacizumab combination will be given every 21 days, atezolizumab 1200 mg and bevacizumab 15 mg/kg will be administered intravenously on a Q3 week schedule.
  Subjects will start the combination of bevacizumab and atezolizumab followed by TACE treatment 4 weeks ±1 week or up to 5 weeks after study drugs. Full recovery from the procedure is required prior to systemic treatment.
  Interventions: Drug: Atezolizumab Injection; Drug: Bevacizumab; Combination Product: Transarterial chemoembolization

INTERVENTIONS:
Drug: Atezolizumab Injection — Atezolizumab is a monoclonal antibody medication used to treat urothelial carcinoma, non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), small cell lung cancer (SCLC), hepatocellular carcinoma, and alveolar soft part sarcoma It is a fully humanized, engineered monoclonal antibody of Immunoglobulin G1 (IgG1) isotype against the protein programmed cell death-ligand 1 (PD-L1).
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab, is a medication used to treat a number of types of cancers and a specific eye disease. For cancer, it is given by slow injection into a vein (intravenous) and used for colon cancer, lung cancer, glioblastoma, and renal-cell carcinoma. In many of these diseases it is used as a first-line therapy. For age-related macular degeneration it is given by injection into the eye (intravitreal).
  Other Names: Avastin
Combination Product: Transarterial chemoembolization — Transarterial chemoembolization (TACE) is a local therapy for HCC which induces tumor necrosis.
  Other Names: TACE

SUMMARY:
There is an unmet need for patients with intermediate stage hepatocellular carcinoma (HCC). It is known that local tumor ablation can increase tumor immunogenicity by releasing tumor associated antigens, potentially increasing the response to immune therapy not just locally, but systemically. In addition, there is now positive data with immune therapy in advanced HCC, there is renewed interest in the combination of local therapy and systemic therapy in Barcelona Clinic Liver Clinic B (BCLC B) patients with systemic therapies other than sorafenib. Based on this data, the investigators plan to examine the atezolizumab and bevacizumab combination with Transarterial Chemoembolization (TACE) in patients with BCLC B HCC.

DETAILED DESCRIPTION:
Targeting the Programmed Death-Ligand 1 (PD-L1) pathway with atezolizumab has demonstrated activity in patients with advanced malignancies who have failed standard-of-care therapies. Objective responses have been observed across a broad range of malignancies, including Non-Small-Cell Lung Cancer (NSCLC), urothelial carcinoma, Renal Cell Carcinoma (RCC), melanoma, colorectal cancer, head and neck cancer, gastric cancer, breast cancer, and sarcoma (see Atezolizumab Investigator's Brochure for detailed efficacy results).

Atezolizumab has been generally well tolerated. Adverse events with potentially immune-related causes consistent with an immunotherapeutic agent, including rash, influenza-like illness endocrinopathies, hepatitis or transaminitis, pneumonitis colitis, and myasthenia gravis, have been observed (see Atezolizumab Investigator's Brochure for detailed safety results). To date, these events have been manageable with treatment or interruption of atezolizumab treatment.

The combination of atezolizumab and bevacizumab in HCC has been well studied in both the phase 1 G030140 study and the phase 3 IMBrave150 study with response rates of 36% and 27% respectively. A phase 2 study of bevacizumab and TACE showed that the combination can be safely administered on the same day. Given concern for risk of bleeding with bevacizumab, all patients on these two studies had recent Endoscopic Gastroduodenoscopies (EGDs) and no patients with untreated varices were included. The risk of bleeding on both studies were reported as low, and risk of benefit was presented as outweighing risk.

This trial will enroll patients with HCC who have BCLC B disease and are not candidates for curative treatment but are candidates for TACE. Typically, these patients would be treated with local treatment alone, but given the relatively poor prognosis and limited treatment options for these patients, this population is considered appropriate for trials of novel therapeutic candidates. The benefit-risk ratio for atezolizumab and bevacizumab in combination with TACE is expected to be acceptable in this setting.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 within 28 days prior to registration
* No cirrhosis or Child-Pugh A cirrhosis
* Diagnosis of HCC either by imaging or biopsy
* Evidence of HCC that meets BCLC B criteria
* Patients must have adequate hepatic, bone marrow, and renal function. All screening labs should be performed within 14 days of treatment initiation.
* Patients must be candidates for TACE treatment that can be treated in up to 4 sessions
* Patients who are positive for Hepatitis B (HBc), regardless of HBs status, and have an undetectable Hepatitis B virus (HBV) viral load do not require HBV antiviral prophylaxis
* Patients who are not on HBV therapy, but positive for Hepatitis B surface antigen (HBsAg) and have an undetectable viral load are eligible for the study as long as they begin anti-viral prophylaxis prior to the start of study treatment
* Patients can have untreated hepatitis C
* At least one unidimensional tumor measurable by RECIST v1.1 criteria
* Hg ≥ 9 g/dL
* Creatinine less than 1.5 x ULN
* Serum bilirubin < 2.5 mg/dl
* Aspartate Transferase (AST) < 5X upper limit of normal (ULN)
* Alanine Transaminase (ALT) < 5X ULN
* Platelet count > 100 x 10^9/L
* Patients must have an EGD within 6 months with no evidence of esophageal and/or gastric varices with bleeding or high risk of bleeding. Patients with varices must be assessed and treated per local standard-of-care prior to enrollment.
* Ability to comply with the study protocol, in the investigator's judgment
* Life expectancy ≥ 6 months
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:
* Absolute Neutrophil Count (ANC) ≥1.5 · 10^9/L (1500/ÍL) without granulocyte colony-stimulating factor support
* Lymphocyte count ≥ 0.5 ∙ 10^9/L (500/ÍL)
* Serum albumin ≥ 25 g/L (2.5 g/dL)
* For patients not receiving therapeutic anticoagulation: International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 ∙ ULN
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen allowed for both Atezo and Avastin. Please note the most current guidelines for Avastin are: Exclusionary: Current or recent (< 10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day), or clopidogrel (> 75 mg/day) Allowed: Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or aPTT is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for ≥ 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below. Women of child-bearing potential must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of atezolizumab and bevacizumab. Women must refrain from donating eggs during this same period.

  1. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  2. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
* For men of childbearing potential: With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of atezolizumab and bevacizumab to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure.

Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible

Exclusion Criteria:

* Patients must not have signs of liver failure or history of liver failure e.g. - encephalopathy or variceal bleeding
* Uncontrolled hepatitis B infection with viral load >500 IU/ml
* History of hypertensive crisis or hypertensive encephalopathy
* Patients who are candidates for curative intent therapy (transplant, resection, or thermal ablation) or liver transplant
* Patients who are on the transplant list
* Ascites requiring therapeutic paracentesis in the last 12 months
* Episode of hepatic encephalopathy in the last 12 months
* Extrahepatic spread: borderline portal lymph nodes deemed to be of indeterminate nature and measuring less than 2 cm are allowed
* Prior local or systemic therapy for HCC or prior TACE, excluding prior use of Radiofrequency Ablation (RFA)
* Patients cannot have known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Occlusion of the hepatic artery or main portal vein
* Pregnant or lactating, or intending to become pregnant during the study
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or other recombinant human antibodies
* Known history of Human Immunodeficiency virus (HIV) infection. No HIV testing is required.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 8 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

  1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  i. Rash must cover < 10% of body surface area ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of leptomeningeal disease
* Active tuberculosis
* Uncontrolled tumor-related pain

  a. Patients requiring pain medication must be on a stable regimen at study entry.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Signs or symptoms of significant infection within 2 weeks prior to Day 1
* Severe infection within 4 weeks prior to initiation of study treatment, including but not limited hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Received therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1, Day 1
* Significant cardiovascular disease, (such as New York Heart Association cardiac disease Class II or greater, myocardial infarction, or cerebrovascular accident) within 3 months prior to prior to Day 1, unstable arrhythmias, or unstable angina
* Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* History of stroke, prolonged reversible ischemic neurological deficit or transient ischemic attack within 6 months prior to Day 1
* Major surgical procedure within 28 days prior to Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Live, attenuated vaccines (e.g., FluMist®) are prohibited within 4 weeks prior to initiation of study treatment, during treatment with atezolizumab, and for 5 months after the last dose of atezolizumab.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Malignancies within 2 years prior to study start, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year Overall Survival (OS) > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  a. Patients with indwelling catheters (e.g., PleurX®) are allowed.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure [BP] ≥150 mmHg and/or diastolic BP >100 mmHg), based on an average of ≥ 3 BP readings on ≥ 2 sessions. Anti-hypertensive therapy to achieve these parameters is allowable
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy
* Current or recent (within 10 days of first dose of study treatment) use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
* Current or recent (< 10 days prior to initiation of study treatment) use of aspirin (> 325 mg/day), or clopidogrel (> 75 mg/day) Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or aPTT is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for ≥ 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days of treatment start
* Proteinuria, as demonstrated by urine dipstick or ≥1.0 g of protein in a 24-hour urine collection. All patients with ≥2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein.
* Chronic daily treatment with a nonsteroidal anti-inflammatory drug (occasional use for the symptomatic relief of medical conditions such as headache or fever is allowed)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti- cytotoxic T-lymphocyte associated protein 4 (CTLA-4), anti- Programmed cell death protein 1 (PD-1), and anti- Programmed death-ligand 1 (PD-L1) therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the bevacizumab or atezolizumab formulation
* History of Grade ≥ 4 venous thromboembolism
* History of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess, or active GI bleeding within 6 months prior to randomization
* Serious, non-healing wound, active ulcer, or untreated bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Stein, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adashek ML, Feldman M. Cytokine Release Syndrome Resulting From Anti-Programmed Death-1 Antibody: Raising Awareness Among Community Oncologists. J Oncol Pract. 2019 Sep;15(9):502-504. doi: 10.1200/JOP.19.00160. Epub 2019 Jul 16. No abstract available. PMID 31310573
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Ravelli A, Minoia F, Davi S, Horne A, Bovis F, Pistorio A, Arico M, Avcin T, Behrens EM, De Benedetti F, Filipovic L, Grom AA, Henter JI, Ilowite NT, Jordan MB, Khubchandani R, Kitoh T, Lehmberg K, Lovell DJ, Miettunen P, Nichols KE, Ozen S, Pachlopnik Schmid J, Ramanan AV, Russo R, Schneider R, Sterba G, Uziel Y, Wallace C, Wouters C, Wulffraat N, Demirkaya E, Brunner HI, Martini A, Ruperto N, Cron RQ; Paediatric Rheumatology International Trials Organisation; Childhood Arthritis and Rheumatology Research Alliance; Pediatric Rheumatology Collaborative Study Group; Histiocyte Society. 2016 Classification Criteria for Macrophage Activation Syndrome Complicating Systemic Juvenile Idiopathic Arthritis: A European League Against Rheumatism/American College of Rheumatology/Paediatric Rheumatology International Trials Organisation Collaborative Initiative. Arthritis Rheumatol. 2016 Mar;68(3):566-76. doi: 10.1002/art.39332. Epub 2016 Feb 9. PMID 26314788
- [Background] Riegler LL, Jones GP, Lee DW. Current approaches in the grading and management of cytokine release syndrome after chimeric antigen receptor T-cell therapy. Ther Clin Risk Manag. 2019 Feb 28;15:323-335. doi: 10.2147/TCRM.S150524. eCollection 2019. PMID 30880998
- [Background] Rotz SJ, Leino D, Szabo S, Mangino JL, Turpin BK, Pressey JG. Severe cytokine release syndrome in a patient receiving PD-1-directed therapy. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26642. Epub 2017 May 24. PMID 28544595
- [Background] Schram AM, Berliner N. How I treat hemophagocytic lymphohistiocytosis in the adult patient. Blood. 2015 May 7;125(19):2908-14. doi: 10.1182/blood-2015-01-551622. Epub 2015 Mar 10. PMID 25758828
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- See also: Clinical features and diagnosis of hemophagocytic lymphohistiocytosis — https://www.uptodate.com/contents/clinical-features-and-diagnosis-of-hemophagocytic-lymphohistiocytosis

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab and Bevacizumab in Combination With TACE: THIS IS A SINGLE ARM PILOT/FEASIBILITY STUDY. THE STUDY CONSISTS OF A SCREENING PERIOD (DAY -28 TO DAY -1), A TREATMENT PERIOD, AND A TREATMENT DISCONTINUATION VISIT.
  The atezolizumab and bevacizumab combination will be given every 21 days, atezolizumab 1200 mg and bevacizumab 15 mg/kg will be administered intravenously on a Q3 week schedule.
  Subjects will start the combination of bevacizumab and atezolizumab followed by TACE treatment 4 weeks ±1 week or up to 5 weeks after study drugs. Full recovery from the procedure is required prior to systemic treatment.
  For cancer, it is given by slow injection into a vein (intravenous) and used for colon cancer, lung cancer, glioblastoma, and renal-cell carcinoma. In many of these diseases it is used as a first-line therapy. For age-related macular degeneration it is given by injection into the eye (intravitreal).
  Transarterial chemoembolization: Transarterial chemoembolization (TACE) is a local therapy for HCC which induces tumor necrosis.
Period: Overall Study
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or Higher Treatment Related Adverse Events
Description: Safety and tolerability will be assessed by the rate of grade 3 or higher Adverse Events (AEs), graded using the CTCAE version 5. The rate will be assessed using the Bayesian Predictive Probability approach. Due to early termination of the study, reported here is the number of participants that experienced any grade 3 or higher event.
Time Frame: up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Response Rate in Solid Tumors
Description: Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) will be used to assess overall response rate. Complete Response (CR): disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD). Due to early termination of the study, a formal overall response rate could not be calculated. Presented here is the overall response frequency by RECIST 1.1 criteria type.
Time Frame: up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 3
Participants
  Partial response (PR) | 0
  Stable disease (SD) | 0
  Complete Response (CR) | 3
  Progressive Disease (PD) | 0

3. Secondary Outcome: Response Rate in Hepatocellular Carcinoma
Description: Response Evaluation Criteria in Hepatocellular Carcinoma-Specific Modified RECIST (HCC mRECIST) will be used to assess overall response rate. Complete response (CR): When all visible tumor areas on the arterial phase disappear, indicating complete necrosis. Partial response (PR): A significant decrease (≥ 30%) in the size of the enhancing tumor areas on the arterial phase. Stable disease (SD): No significant change in tumor size, neither shrinkage nor progression. Progressive disease (PD): An increase in the size of the enhancing tumor areas on the arterial phase (≥ 20%) or the appearance of new enhancing lesions.
Time Frame: up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 3
Participants
  Partial Response (PR) | 0
  Stable Disease (SD) | 0
  Complete Response (CR) | 3
  Progressive disease (PD) | 0

4. Secondary Outcome: Time to Progression
Description: Defined as the time from trial enrollment until objective tumor progression by RECIST, Response Evaluation Criteria in Solid Tumors criteria.
Time Frame: up to 18 months
Population: Data not collected.
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to TACE Progression (TTTP)
Description: Defined as the interval of time from the day of the images after a TACE procedure to the time or progression, new vascular invasion or extrahepatic spread also is counted as progression.
Time Frame: up to 18 months
Population: Data not collected.
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Untaceable Progression
Description: Defined as time to untreatable tumor progression and/or transient deterioration to Child-Pugh C score and/or appearance of vascular invasion/extrahepatic spread. Child-Pugh score ranges from 5-15. Child-Pugh C = 10-15. A higher score indicates a worse outcome.
Time Frame: up to 18 months
Population: Data not collected.
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Atezolizumab and Bevacizumab in Combination With TACE: THIS IS A SINGLE ARM PILOT/FEASABILITY STUDY. THE STUDY CONSISTS OF A SCREENING PERIOD (DAY -28 TO DAY -1), A TREATMENT PERIOD, AND A TREATMENT DISCONTINUATION VISIT.
  The atezolizumab and bevacizumab combination will be given every 21 days, atezolizumab 1200 mg and bevacizumab 15 mg/kg will be administered intravenously on a Q3 week schedule.
  Subjects will start the combination of bevacizumab and atezolizumab followed by TACE treatment 4 weeks ±1 week or up to 5 weeks after study drugs. Full recovery from the procedure is required prior to systemic treatment.
  For cancer, it is given by slow injection into a vein (intravenous) and used for colon cancer, lung cancer, glioblastoma, and renal-cell carcinoma. In many of these diseases it is used as a first-line therapy. For age-related macular degeneration it is given by injection into the eye (intravitreal).
  Transarterial chemoembolization: Transarterial chemoembolization (TACE) is a local therapy for HCC which induces tumor necrosis.
Arm/Group | Atezolizumab and Bevacizumab in Combination With TACE
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab and Bevacizumab in Combination With TACE (N=3)
Fatigue (General disorders) | 2
Edema limbs (General disorders) | 1
Flu like symptoms (General disorders) | 1
Pain (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05776875/Prot_SAP_000.pdf